CLINICAL TRIAL: NCT05684497
Title: Low Back Pain Support Program During Pregnancy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Munevver Aybuke Berber Cikrik, Assistant professor, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Kastamonu University
Record Dates: First submitted 2022-01-16; First posted 2023-01-13 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain; Pregnancy Related; Nurse's Role
Keywords: Back Pain; Life Quality; Nursing; Pregnancy, Pender's Health Promotion Model
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The intervention group was conducted a LBPSP
  Interventions: Behavioral: LBPSP in Pregnancy
- control group (No Intervention): the control group were not and were left to routine antenatal care.

INTERVENTIONS:
Behavioral: LBPSP in Pregnancy — LBPSP is a 50-minute interactive presentation as face to face program according to Pender's Health Promotion Model Parameters.
  Arms: experimental group

SUMMARY:
Purpose of Research: The study was conducted as a randomized controlled experimental study to evaluate the effect of the Low Back Pain During Pregnancy Support Program (LBPSP).

Research Hypotheses H1: The perception of back pain during pregnancy in the intervention group receiving the "Low Back Pain During Pregnancy Support Program (LBPSP) will decrease compared to the control group.

H2: The Oswestry Disability Index scores of the intervention group receiving the Low Back Pain During Pregnancy Support Program (LBPSP) will decrease compared to the control group.

First interview Introductory Information Form, Low Back Pain Evaluation Form, Visual Analog Scale (VAS), and Oswestry Disability Index were applied to all pregnant women in the intervention and control groups participating in the study as pre-test at the first interview. The intervention group was conducted a LBPSP, the control group were not and were left to routine antenatal care.Four weeks after the first interview, Intervention and control groups were interviewed again, and the Low Back Pain Evaluation Form and Oswestry Disability Index scales were applied. In addition, the LBPSP Evaluation Form prepared by the researcher was applied to the pregnant women in the intervention group to evaluate the LBPSP.

DETAILED DESCRIPTION:
The research population consisted of all pregnant women registered at a Family Health Center between July 2021 and July 2022.The power of the study was calculated in the G*Power (v3.1.9.4) program to determine the number of samples. Oswestry Disability Index was taken as the main parameter in the study. In the survey conducted by Pekcetin et al., the Oswestry Disability Index scale score average of the group to be trained was found to be 39.53 ±14.04 before the training and 26.96 ±13.69 after the training (Pekcetin et al., 2019). In the statistical analysis performed by taking the results of this study as a criterion, the alpha reliability level of the survey was taken as 0.01. The power was 80%, and according to the Oswestry Disability Index scale, the score was average. It was determined that 36 pregnant women should be included in the group. However, considering the possibility of data loss, a total of 80 pregnant women, 40 were included in the group that would be included in the low back pain prevention and coping support program in addition to routine pregnant care, and 40 were included in the group that would receive only routine antenatal care.

The allocation of intervention and control groups was determined using the simple random sampling method (random.org). The numbers determined by the simple random sampling method became the appointment order.

Criteria for inclusion in the study;

* Read and write in Turkish,
* 18 years and over aged,
* Three or more score low back pain according to VAS
* Singleton pregnancy

Exclusion criteria from the study:

* Gynecological or urological problems that cause pain during pregnancy (premature birth, pyelonephritis, etc.)
* Using analgesics during pregnancy,
* Risky pregnancies for which bed rest is recommended during pregnancy,
* Were not included in the study. After the researcher called the pregnant women via phone and evaluated their compliance with the research criteria, the pregnant women who met the inclusion criteria were informed about the research and invited to the study. Data were collected by face-to-face interviews with all pregnant women in the study in an isolated room.

First interview Introductory Information Form, Low Back Pain Evaluation Form, Visual Analog Scale (VAS), and Oswestry Disability Index were applied to all pregnant women in the intervention and control groups participating in the study as pre-test at the first interview. The intervention group was conducted a LBPSP, the control group were not and were left to routine antenatal care.Four weeks after the first interview, Intervention and control groups were interviewed again, and the Low Back Pain Evaluation Form and Oswestry Disability Index scales were applied. In addition, the LBPSP Evaluation Form prepared by the researcher was applied to the pregnant women in the intervention group to evaluate the LBPSP.

The purpose and content of LBPSP was explained and contucted to the intervention group. LBPSP is a 50-minute interactive presentation as face to face program according to Pender's Health Promotion Model Parameters. LBPSP content is given in Figure 3. And also, a special LBPSP handbook has been prepared for this program, enriched with visuals for pregnant women and printed. This handbook was given to the intervention group after LBPSP.

ELIGIBILITY:
Inclusion criteria

* Read and write in Turkish,
* 18 years and over aged,
* Three or more score low back pain according to VAS
* Singleton pregnancy

Exclusion Criteria:

Gynecological or urological problems that cause pain during pregnancy (premature birth, pyelonephritis, etc.)

* Using analgesics during pregnancy,
* Risky pregnancies for which bed rest is recommended during pregnancy,
* Were not included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
pregnancy related low back pain | each participant will be re-evaluated at the end of 4 weeks
  measurement of low back pain life status of pregnant women with VAS
quality of life in pregnancy | each participant will be re-evaluated at the end of 4 weeks
  measurement of pregnant women's quality of life with Oswestry disability index

CONTACTS AND LOCATIONS:
Overall Officials: Münevver Aybüke Berber Çıkrık, Study Director — Istanbul University Cerrahpasa Institute of Graduate Education Studies; Münevver Aybüke Berber Çıkrık, Study Director — stanbul University Cerrahpasa Institute of Graduate Education Studies
Locations (1):
- Münevver Aybüke Berber Çıkrık, Kastamonu, Kastamonu/Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No